CLINICAL TRIAL: NCT07403370
Title: Olanzapine 2.5 mg Versus 5 mg Versus 10 mg in Highly Emetogenic Regimens: A Systematic Review and Network Meta-Analysis of Randomized Controlled Trials.
Brief Title: Olanzapine Dose Comparison for the Prevention of HER-INV: A Network Meta-Analysis
Status: Recruiting | Type: Observational
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Fangchao Zheng, MD, Clinical associate professor, Shandong Cancer Hospital and Institute
Other Study IDs: SDTHEC-IF
Record Dates: First submitted 2026-01-18; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumours; Olanzapine; Nausea and Vomiting
Keywords: Olanzapine; Network Meta-Analysis; High emetic risk; Nausea and Vomiting; Solid tumours
MeSH Terms: conditions — Nausea; Vomiting | interventions — Olanzapine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Olanzapine Doses 2.5mg
  Interventions: Drug: Olanzapine (dose comparison: 2.5 mg, 5 mg, 10 mg)
- Olanzapine Doses 5mg
  Interventions: Drug: Olanzapine (dose comparison: 2.5 mg, 5 mg, 10 mg)
- Olanzapine Doses 10mg
  Interventions: Drug: Olanzapine (dose comparison: 2.5 mg, 5 mg, 10 mg)

INTERVENTIONS:
Drug: Olanzapine (dose comparison: 2.5 mg, 5 mg, 10 mg) — Olanzapine (dose: 2.5 mg) vs. olanzapine (dose: 5 mg) vs. olanzapine (dose: 10 mg)

SUMMARY:
Olanzapine is an effective antiemetic agent for preventing highly emetogenic regimens-induced nausea and vomiting (HER-INV) in patients receiving highly emetogenic regimens (HER). The optimal dose remains debated, with the standard 10 mg dose often causing significant daytime sedation. Recent evidence suggests that lower doses (2.5 mg and 5 mg) may offer comparable efficacy with improved tolerability. However, no head-to-head randomized controlled trials (RCTs) directly compare all three doses.

DETAILED DESCRIPTION:
To compare the relative efficacy and safety of olanzapine at 2.5 mg, 5 mg, and 10 mg, in combination with standard triple antiemetic prophylaxis, for the prevention of HER-INV in adult patients undergoing HER, using a network meta-analysis (NMA) of RCTs. RCTs comparing any two doses of olanzapine (2.5 mg, 5 mg, 10 mg) in adults with solid tumors.

Inclusion Criteria:

1. Olanzapine was used to prevent nausea and vomiting (HER-INV) in solid tumors patients receiving highly emetogenic regimens
2. Randomized controlled trials (RCTs), including conference abstracts if sufficient data are provided.
3. Adult patients (≥18 years) with solid tumors receiving highly emetogenic chemotherapy (HEC).

3. Olanzapine at 2.5 mg, 5 mg, or 10 mg, added to a standard triple antiemetic regimen (NK1 receptor antagonist + 5-HT3 receptor antagonist + dexamethasone).

4. Any of the other three olanzapine doses or placebo (2.5 mg vs. 5 mg vs. 10 mg, or vs. placebo).

5. At least one of the pre-specified efficacy or safety outcomes must be reported.

Exclusion Criteria:

1. Non-solid tumors patients, non-randomized studies, observational studies, case reports, reviews.
2. Studies involving pediatric populations, non-HEC regimens.
3. Studies where olanzapine is used as rescue medication only.
4. Studies with overlapping patient populations (the most recent or complete publication will be selected).

Information Sources: Electronic databases: PubMed, Embase, Cochrane Central Register of Controlled Trials (CENTRAL), Web of Science Core Collection. We will also search clinical trial registries (ClinicalTrials.gov, WHO ICTRP) and manually review reference lists of relevant systematic reviews and included studies.

Risk of Bias Assessment: The risk of bias for individual RCTs will be assessed using the revised Cochrane Risk of Bias tool for randomized trials (RoB 2.0) by two independent reviewers.

Subgroup Analyses: Subgroup analyses are planned by treatment regimens (such as: cisplatin-based vs. AC-based et al.).

ELIGIBILITY:
Inclusion Criteria:

1. Olanzapine was used to prevent nausea and vomiting (HER-INV) in solid tumors patients receiving highly emetogenic regimens.
2. Randomized controlled trials (RCTs), including conference abstracts if sufficient data are provided.
3. Adult patients (≥18 years) with solid tumors receiving highly emetogenic chemotherapy (HEC).

3. Olanzapine at 2.5 mg, 5 mg, or 10 mg, added to a standard triple antiemetic regimen (NK1 receptor antagonist + 5-HT3 receptor antagonist + dexamethasone).

4. Any of the other three olanzapine doses or placebo (2.5 mg vs. 5 mg vs. 10 mg, or vs. placebo).

5. At least one of the pre-specified efficacy or safety outcomes must be reported.

Exclusion Criteria:

1. Non-solid tumors patients, non-randomized studies, observational studies, case reports, reviews.
2. Studies involving pediatric populations, non-HEC regimens.
3. Studies where olanzapine is used as rescue medication only. Studies with overlapping patient populations (the most recent or complete publication will be selected).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with solid tumors received different doses of olanzapine (2.5 mg, 5 mg, 10 mg) as an add-on to standard antiemetic prophylaxis for the prevention of HER-induced nausea and vomiting in adult (≥18 years) patients with solid tumors receiving highly emetogenic regimens.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-18 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The complete response rate of nausea and vomiting in the overall phase (including acuted and delayed phase) by highly emetogenic regimens in solid tummors. | Nausea and vomiting complete response was assesed during the treatment period (or during the overall assessment period) after the initiation of highly emetogenic regimens, up to 4 weeks.
  Nausea and vomiting complete response (CR; no vomiting or retching, no rescue medication) rate in the overall phase (including acuted [0-24h] and delayed [>24h] phase ) after highly emetogenic regimens in solid tummors .

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No